CLINICAL TRIAL: NCT05359159
Title: Follow-up of Patients With Previous SARS-CoV-2 Infection: Long-term Damage Assessment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Clara Balsano, Full professor, University of L'Aquila
Other Study IDs: 66848
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: COVID-19
Keywords: Long-COVID; post-COVID; SarS-CoV2
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-COVID patients: Patients recovered from Sars-CoV2 infection
  Interventions: Other: Data collection
- healthy control patients: Patients who did not have Sars-CoV2
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collection

SUMMARY:
People affected by SARS-CoV-2 infection, whether patients have developed mild forms or a severe form of the disease, complain of nonspecific and entirely new symptoms or complain about the persistence pf them.Investigators intend to follow over time the post-infectious phase of patients discharged from sub-intensive care unit. The aim is to identify symptoms and their frequency of presentation in the SARS-CoV-2 population in the post-acute period.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18

Exclusion Criteria:

* Patients under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients admitted to Ospedale San Salvatore dell'Aquila over 18 years during Sars-CoV2 pandemics, with or without Sars-CoV2 related disease
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Greater understanding of SARS-CoV-2 disease | 24 months
  Greater understanding of SARS-CoV-2 disease and its long-term manifestations. To this end, the clinical manifestations, any alterations in laboratory and instrumental parameters will be evaluated to identify organ damages and calculate its prevalence

SECONDARY OUTCOMES:
Measurement of psychological impact of SARS-CoV-2 disease | 24 months
  Understanding the impact of the disease and its sequelae on daily life and the impact on the psychological aspect of the person;

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Clara Balsano, L’Aquila, Italy/L'Aquila
  - University of L'Aquila, L’Aquila